CLINICAL TRIAL: NCT01995682
Title: Evaluate the Feasibility of the NLA Tool, a Combined Assessment of Nutritional and Physical Functional Status, to Provide Personalized Advice for the Independence and Mobility of Elderly
Brief Title: Feasibility Clinical Study of NLA Tool-US
Acronym: NLA
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 12.34.NRC
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Independent living; walk with or without walking aids

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens are to be collected or retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is to evaluate the feasibility of the NLA tool, a combined assessment of nutritional and physical functional status, to provide personalized advice for the independence and mobility of elderly.

DETAILED DESCRIPTION:
* Determining the proportion of elderly subjects who, according to the NLA result, would qualify for a personalized program to improve their nutritional and physical status;
* Determining the segmentation (defined by cut-off criteria) of these elderly subjects stratified into 3 NLA subgroups according to strength and endurance performance (33% +/- 10% of target group)

ELIGIBILITY:
Inclusion Criteria:

1. aged between 65 and 90 years,
2. able to walk with or without walking aid,
3. having obtained the subject's written informed consent
4. free of cognitive impairment (3MSE),

Exclusion Criteria:

1. self reported restriction to exercise(by a physician or other).
2. unable to carry out performance tests and questionnaires correctly,
3. self reported lower or upper extremity surgery or fracture in the last 3 months
4. self-reported symptomatic coronary artery disease, myocardial infarction in last 6 months
5. self reported history of neurological disease (e.g., Parkinson disease, stroke) with residual impairment
6. uncontrolled hypertension (>150/90 mm Hg)
7. self reported congestive heart failure
8. unable to communicate in English. Non-English speaking individuals will be excluded due to safety concerns in being able to understand testing instructions.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Independently living men and women at 65-90 years old who are able to walk with or without walking aid
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
NLA feasibility | One day
  Determining the proportion of elderly subjects who, according to the NLA result, would qualify for a personalized program to improve their nutritional and physical status.

SECONDARY OUTCOMES:
Evaluate the average time required for completing the NLA | One day
  Measure the time required to complete the NLA.

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Fielding, Ph.D., Principal Investigator — Jean Mayer USDA Human Nutrition Research Center on Aging, Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts, United States